CLINICAL TRIAL: NCT05945563
Title: Clopidogrel Hyper-Responsiveness: Incidence and Associated Outcomes in Patients With Cerebral Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 120.VAS.2022.D
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry study will investigate the incidence of and outcomes associated with clopidogrel hyper-responsive patients treated at Methodist Dallas Medical Center, beginning in January 2018, who suffered cerebral aneurysms.

DETAILED DESCRIPTION:
This registry study will investigate the incidence of and outcomes associated with clopidogrel hyper-responsive patients treated at Methodist Dallas Medical Center, beginning in January 2018, who suffered cerebral aneurysms.

Perioperative and short-term clinical data will be obtained from electronic medical records. All the data variables will be documented in an Excel sheet (Appendix B). This section will provide an overview of the data collected which will include, but are not limited to, the following:

• Pre-Operative Information: Demographics (e.g., age, gender), patient characteristics (e.g., BMI, American Society of Anesthesiologists class), and pre-operative medical history (e.g., tobacco use; comorbidities: hypertension, cardiopulmonary disease, diabetes; etc.).

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older Diagnosed with cerebral aneurysms (i.e. ICD-10 i67.1) Pre-intervention treatment with clopidogrel

Exclusion Criteria:

* Does not meet inclusion criteria specified in 3.1

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and Male age 18 or older
Study Population: Age 18 years or older Diagnosed with cerebral aneurysms (i.e. ICD-10 i67.1) Pre-intervention treatment with clopidogrel
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
Registry Evaluation | 90 days
  The demographic characteristics, treatment strategies, incidence, and outcomes in patients hyper-responsive to clopidogrel.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Smith SC Jr, Feldman TE, Hirshfeld JW Jr, Jacobs AK, Kern MJ, King SB 3rd, Morrison DA, O'Neil WW, Schaff HV, Whitlow PL, Williams DO, Antman EM, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; ACC/AHA/SCAI Writing Committee to Update 2001 Guidelines for Percutaneous Coronary Intervention. ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/SCAI Writing Committee to Update 2001 Guidelines for Percutaneous Coronary Intervention). Circulation. 2006 Feb 21;113(7):e166-286. doi: 10.1161/CIRCULATIONAHA.106.173220. No abstract available. PMID 16490830
- [Background] O'Donoghue M, Wiviott SD. Clopidogrel response variability and future therapies: clopidogrel: does one size fit all? Circulation. 2006 Nov 28;114(22):e600-6. doi: 10.1161/CIRCULATIONAHA.106.643171. No abstract available. PMID 17130347
- [Background] Damman P, Woudstra P, Kuijt WJ, de Winter RJ, James SK. P2Y12 platelet inhibition in clinical practice. J Thromb Thrombolysis. 2012 Feb;33(2):143-53. doi: 10.1007/s11239-011-0667-5. PMID 22183178
- [Background] Jaremo P, Lindahl TL, Fransson SG, Richter A. Individual variations of platelet inhibition after loading doses of clopidogrel. J Intern Med. 2002 Sep;252(3):233-8. doi: 10.1046/j.1365-2796.2002.01027.x. PMID 12270003
- [Background] Muller I, Besta F, Schulz C, Massberg S, Schonig A, Gawaz M. Prevalence of clopidogrel non-responders among patients with stable angina pectoris scheduled for elective coronary stent placement. Thromb Haemost. 2003 May;89(5):783-7. PMID 12719773
- [Background] Serebruany VL, Steinhubl SR, Berger PB, Malinin AI, Bhatt DL, Topol EJ. Variability in platelet responsiveness to clopidogrel among 544 individuals. J Am Coll Cardiol. 2005 Jan 18;45(2):246-51. doi: 10.1016/j.jacc.2004.09.067. PMID 15653023